CLINICAL TRIAL: NCT02178124
Title: A Phase I Clinical Study, Randomized, Single-blind, Placebo-controlled, Multiple Doses, Dose Escalation Study of the Safety, Tolerability and Pharmacokinetics of Donepezil Patch in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icure Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IPI-002
Record Dates: First submitted 2014-06-27; First posted 2014-06-30 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- dosage 1 (Experimental): drug : 9 people(87.5mg/25cm2) placebo : 3 people(0mg/25cm2)
  Interventions: Drug: Donepezil; Drug: placebo
- dosage 2 (Experimental): dosage2 period 1 : oral administration drug : 12 people(10mg)
  dosage 2 period 2: transdermal administration drug : 9 people(175mg/50cm2) placebo : 3 people(0mg/50cm2)
  Interventions: Drug: Donepezil; Drug: placebo

INTERVENTIONS:
Drug: Donepezil
Drug: placebo

SUMMARY:
Study of the Safety, tolerability and pharmacokinetics with multiple doses of donepezil patch in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* BMI : more than 19 ㎏/㎡, less than 27 ㎏/㎡
* Systolic blood pressure : more than 90, less than 140 (mmHg)
* Diastolic blood pressure : more than 60, less than 100 (mmHg)

Exclusion Criteria:

* Evidence of clinically significant, severe, active, or unstable gastrointestinal, renal,hepatic, respiratory, hematological, endocrine, or cardiovascular system disease.
* A history of skin disease or skin graft
* Hypersensitivity to donepezil or piperidine derivatives or any of the excipients.
* A known or suspected history of drug or alcohol dependency or abuse
* Patients who have participated in another clinical study within 60 days.
* Whole blood within 60 days, apheresis within 30 days, transfusion within 30 days
* Heavy alcohol intake(more than 21 units/week)
* Heavy smoker(more than 10 cigarette/day)
* Abnormal clinical laboratory values which are judged clinically significant by the investigator.
* Any condition that would make the patient or the caregiver, in the opinion of the investigator, unsuitable for the study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
safety and tolerability evaluation | patch : -1d~33d, oral : -1~11d
  evaluation item
  1. adverse event
  2. electrocardiographie
  3. vital sign
  4. physical examination
  5. urine, blood test
  6. skin irritation

SECONDARY OUTCOMES:
pharmacokinetics characteristic evaluation | patch: -1~25d, oral -1~11d
  cohort 1
  1d 0h (pre-dose), 4h, 8h, 12h, 24h (2d), 48h (3d), 72h (4d), 144h (7d), 216h (10d), 288h (13d, last dose start), 292h, 296h, 300h, 312h (14d), 336h (15d), 360h (16d, patch removal), 362h, 364h, 368h, 372h, 384h (17d), 408h (18d), 432h (19d), 480h (21d), 528h (23d), 576h (25d)
  cohort 2 1 period Oral Donepezil
  1d 0h (pre-dose), 0.5h, 1h, 1.5h, 2h, 3h, 4h, 8h, 12h, 24h (2d), 48h (3d), 96h (5d), 144h (7d), 192h (9d), 240h (11d)
  period 2 Donepezil Patch: same cohort1
  evaluation item : donepezil conc.
  evaluation variable patch : AUCτ,ss, Cmax,ss, t1/2β, AI (accumulation index), Cav,ss oral : AUClast, AUC0-∞, Cmax, tmax, t1/2β, CL/F

CONTACTS AND LOCATIONS:
Locations (1):
- ASAN Medical Center, Seoul, South Korea